CLINICAL TRIAL: NCT02563158
Title: Short- and Long-term Outcomes of Liver Resection With Versus Without Hepatic Inflow Occlusion for the Hepatitis B Virus-related Hepatocellular Carcinoma: a Prospective Randomized Controlled Trial
Brief Title: Study of Liver Resection With Versus Without Hepatic Inflow Occlusion for the HBV-related HCC
Acronym: OHx-NOHx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Prof. Shichun Lu, Director, Department of Hepatobiliary Surgery, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JFJZYY-GD-15-01; NO. 2012BAI06B01 (Other Grant/Funding Number: National Key Technology R&D Program of China); NO. 2012ZX10002-017 (Other Grant/Funding Number: National S&T Major Project for Infectious Diseases of China)
Record Dates: First submitted 2015-09-26; First posted 2015-09-30 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Liver Cancer; Surgery
Keywords: liver resection; blood inflow control; ischemia-reperfusion injury; inflammatory response; randomized controlled trial
MeSH Terms: conditions — Liver Neoplasms; Reperfusion Injury | interventions — Hepatectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hx with hepatic inflow occlusion (No Intervention): Hepatectomy is carried out using Pringle maneuver in cycles of 15 minutes clamping + 5 minutes unclamping of the hepatoduodenal ligament.
- Hx with non-occlusion technique (Experimental): Hepatectomy without hepatic inflow occlusion (non-occlusion technique)
  Interventions: Procedure: non-occlusion technique

INTERVENTIONS:
Procedure: non-occlusion technique — Hepatectomy is carried out without hepatic inflow control. (non-occlusion technique)
  Other Names: hepatectomy without hepatic inflow occlusion
  Arms: Hx with non-occlusion technique

SUMMARY:
The study aims to compare the perioperative and long-term outcomes of liver resection for HBV-related HCC with versus without hepatic inflow occlusion.

DETAILED DESCRIPTION:
High prevalence of hepatitis B virus (HBV) imposes a huge burden of hepatocellular carcinoma (HCC) in Asia. Liver resection remains the mainstay of treatment for HCC. Hepatic inflow occlusion, known as the Pringle maneuver, is most commonly used to reduce blood loss during liver parenchymal transection. A major issue about this maneuver is the ischemia-reperfusion injury to the remnant liver. And the hemodynamic disturbance to the tumor-bearing liver remains an oncologic concern. Given the technical advances in living donor liver transplantation, vascular occlusion can be avoided in liver resection by experienced hands. This study aims to compare the perioperative and long-term outcomes of liver resection for HBV-related HCC without versus with hepatic inflow occlusion.

This study will include eligible patients with HBV-related HCC elected for liver resection. 57 patients will be enrolled in each randomized arm to detect a 20% difference in the serum level of total bilirubin on postoperative day 5 (80% power and α = 0.05). The secondary endpoints include procedural parameters, perioperative liver function and inflammatory response, postoperative morbidity and mortality, and long-term outcomes. Patients will be followed for up to five years. Data will be statistically analyzed on an intention-to-treat basis.

This prospective randomized controlled trial is designed to evaluate the feasibility of liver resections for HBV-related HCC without vascular occlusion. Clinical implication of its outcomes may change the present surgical practice and fill the oncologic gaps therein.

ELIGIBILITY:
Inclusion Criteria:

1. Elective liver resection due to HBV-related HCC with Barcelona-Clinic Liver Cancer (BCLC) staging 0 or A;
2. Child-Pugh classified A with or without cirrhosis, or reversed to A from B after conventional therapy;
3. Tumors located either in the left or right hemiliver;
4. Resection extent was a hemi-hepatectomy or less;
5. Informed consent.

Exclusion Criteria:

1. Having comorbidity that contraindicates surgery;
2. Participation in concurrent interventional trials with interference to this study;
3. Eligible for laparoscopic hepatectomy;
4. Requiring concomitant procedures, such as digestive, vascular or biliary reconstruction;
5. Lack of compliance for treatment or future follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Serum total bilirubin on postoperative day 5 | 5 days
  Postoperative liver insufficiency characterized by the serum total bilirubin on POD 5.

SECONDARY OUTCOMES:
Intraoperative blood loss | Entire operation duration
  Total blood loss from the incision to the closure of abdomen
Requirement of blood transfusion | Entire operation duration
  The amount of intraoperative blood transfusion
Operative time | Entire operation duration
  The time from induction of anesthesia to the closure of abdomen
Postoperative intensive-care unit (ICU) stay | Duration of stay in ICU
  Duration of stay in ICU
Hospital stay | Duration of hospital stay
  Duration of hospital stay
Total hospital expenditure | Duration of hospital stay
  Total costs during hospital stay
Perioperative systemic inflammatory response | an expected average of 7 days
  Perioperative systemic inflammatory response is characterized by elevated serum level of tumor necrosis factor-α (TNF-α), interleukins (IL)-1α, 2, 6, 8 and 10, procalcitonin (PCT) and C-reactive protein (CRP) at different time points.
Postoperative morbi-mortality | an expected average of 12 days in hospital
  Postoperative morbi-mortality is characterized by postoperative complication and its severity based on Clavien-Dindo classification and in-hospital mortality
Long-term oncologic outcomes | 5 years after operation
  1, 3, 5-year tumor recurrence rate
Long-term survival | 5 years after operation
  1, 3, 5-year overall survival (OS) and disease (tumor)-free survival (DFS)

CONTACTS AND LOCATIONS:
Overall Officials: Shichun Lu, MD, PhD, Principal Investigator — Department of Hepatobiliary Surgery, Chinese PLA General Hospital, 28 Fuxing Road, Haidian, Beijing, 100853, China
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Llovet JM, Fuster J, Bruix J; Barcelona-Clinic Liver Cancer Group. The Barcelona approach: diagnosis, staging, and treatment of hepatocellular carcinoma. Liver Transpl. 2004 Feb;10(2 Suppl 1):S115-20. doi: 10.1002/lt.20034. PMID 14762851
- [Result] Dong JH, Yang SZ, Duan WD, Ji WB, Cai SW, Wang J, Shi XJ, Jiang K, Xia HT, He L, Zhang WZ, Huang XQ, Huang ZQ. [Clinical application of precise liver resection techniques in patients with complicated liver space-occupying lesions]. Zhonghua Wai Ke Za Zhi. 2009 Nov 1;47(21):1610-5. Chinese. PMID 20137393
- [Result] Huang ZQ, Xu LN, Yang T, Zhang WZ, Huang XQ, Liu R, Cai SW, Zhang AQ, Feng YQ, Zhou NX, Dong JH. [Liver resection: single center experiences of 2008 consecutive resections in 20 years]. Zhonghua Wai Ke Za Zhi. 2008 Sep 1;46(17):1314-21. Chinese. PMID 19094562
- [Result] Dong J, Yang S, Zeng J, Cai S, Ji W, Duan W, Zhang A, Ren W, Xu Y, Tan J, Bu X, Zhang N, Wang X, Wang X, Meng X, Jiang K, Gu W, Huang Z. Precision in liver surgery. Semin Liver Dis. 2013 Aug;33(3):189-203. doi: 10.1055/s-0033-1351781. Epub 2013 Aug 13. Danish, English. PMID 23943100
- [Result] Sugiyama Y, Ishizaki Y, Imamura H, Sugo H, Yoshimoto J, Kawasaki S. Effects of intermittent Pringle's manoeuvre on cirrhotic compared with normal liver. Br J Surg. 2010 Jul;97(7):1062-9. doi: 10.1002/bjs.7039. PMID 20632273
- [Result] Kim YI, Song KE, Ryeon HK, Hwang YJ, Yun YK, Lee JW, Chun BY. Enhanced inflammatory cytokine production at ischemia/reperfusion in human liver resection. Hepatogastroenterology. 2002 Jul-Aug;49(46):1077-82. PMID 12143206
- [Result] Katz SC, Shia J, Liau KH, Gonen M, Ruo L, Jarnagin WR, Fong Y, D'Angelica MI, Blumgart LH, Dematteo RP. Operative blood loss independently predicts recurrence and survival after resection of hepatocellular carcinoma. Ann Surg. 2009 Apr;249(4):617-23. doi: 10.1097/SLA.0b013e31819ed22f. PMID 19300227
- [Result] Fu SY, Lau WY, Li GG, Tang QH, Li AJ, Pan ZY, Huang G, Yin L, Wu MC, Lai EC, Zhou WP. A prospective randomized controlled trial to compare Pringle maneuver, hemihepatic vascular inflow occlusion, and main portal vein inflow occlusion in partial hepatectomy. Am J Surg. 2011 Jan;201(1):62-9. doi: 10.1016/j.amjsurg.2009.09.029. Epub 2010 Apr 20. PMID 20409520
- [Derived] Xu Y, Chen J, Wang H, Zheng H, Feng D, Zhang A, Leng J, Duan W, Yang Z, Chen M, Shi X, Cai S, Ji W, Jiang K, Zhang W, Chen Y, Gu W, Dong J, Lu S. Perioperative and long-term outcomes of liver resection for hepatitis B virus-related hepatocellular carcinoma without versus with hepatic inflow occlusion: study protocol for a prospective randomized controlled trial. Trials. 2016 Oct 11;17(1):492. doi: 10.1186/s13063-016-1621-9. PMID 27724929